CLINICAL TRIAL: NCT06898125
Title: Evaluation of Extracorporeal Shockwave Therapy (ESWT) and Complex Decongestive Therapy (CDT) Results in Patients With Lipoedema
Brief Title: Evaluation of Extracorporeal Shockwave Therapy and Complex Decongestive Therapy Results in Patients With Lipedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13.03.2023/16
Record Dates: First submitted 2025-03-18; First posted 2025-03-27 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Lipedema; Pain
Keywords: lipedema; complex decongestive therapy; extracorporeal shockwave therapy
MeSH Terms: conditions — Lipedema; Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: randomized controlled trials
Who Masked: Outcomes Assessor
Masking Description: Outcome measures were assessed by the investigator who was blinded to each patient's group. The participants and therapists were not blinded to the group allocation. Patients were briefed to not disclose which group they were in during the assessment process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complex Decongestive Therapy (Active Comparator): In this group, Complex Decongestive Therapy treatment will be applied to both lower extremities for two weeks, three sessions per week.
  Interventions: Other: Complex Decongestive Therapy
- Extracorporeal Shockwave Therapy (Experimental): This group will receive therapy for two weeks, three sessions per week, with the Modus ESWT® Radial Shockwave Therapy ( İnceler Medikal, Turkey ) brand ESWT device (35mm radial wavy head); 3000 impulse 15 Hz will be applied to both lower extremities with an average energy level of 3.5.
  Interventions: Other: Extracorporeal Shockwave Therapy
- Extracorporeal Shockwave Therapy and Complex Decongestive Therapy (Experimental): In this group, first Extracorporeal Shockwave Therapy and then Complex Decongestive Therapy treatment will be applied in the same session for two weeks, three sessions a week.
  Interventions: Other: Extracorporeal Shockwave Therapy; Other: Complex Decongestive Therapy

INTERVENTIONS:
Other: Extracorporeal Shockwave Therapy — Shock wave therapy is a new modality for the improvement of cellulite and lipedema; it is an easy, noninvasive, local therapy, without side effects, with short periods of application. Its original idea was the stimulation of lipid mobilization and improved lipolysis in areas with edema.
  Arms: Extracorporeal Shockwave Therapy; Extracorporeal Shockwave Therapy and Complex Decongestive Therapy
Other: Complex Decongestive Therapy — Complex decongestive therapy (CDT) is one of the most important treatment modalities of choice for patients with this clinical condition. CDT has two phases: treatment and maintenance. The first stage consists of skin care, manual lymph drainage, kinesiotherapy and bandaging of the limb. Drainage can facilitate the return of lymphatic flow by stimulating the cisterna chyli. Next, kinesiotherapy is applied, which aims to activate the lymph. Finally, the limb is moistened and then a compressive bandage is applied aimed at creating a pressure gradient towards the areas where lymph absorption is greater. The second phase continues skin care, physical exercises and external compression applications using bandages with varying degrees of elasticity.
  Arms: Complex Decongestive Therapy; Extracorporeal Shockwave Therapy and Complex Decongestive Therapy

SUMMARY:
The aim of the study is to evaluate the results of the Extracorporeal Shockwave Therapy and Complex Decongestive Therapy in patient diagnosed with lipedema.

DETAILED DESCRIPTION:
The collected content will be transferred over SPSS 21.0. The normality distribution of the data will be evaluated with the Shapiro-Wilk Test. Data will be displayed as mean±standard deviation, median (1st quartile-3 quartile), or number(percent). In comparisons between the two consuming variables before and after exercise, if the values fit the normal distribution, the "paires sample t test" is used, if not, the Wilcoxon test is used. In the comparison of 3 groups, one-way ANOVA will be applied if it is normally distributed, and if it does not fit the normal distribution, the Kruskal Wallis test will be applied. Post-hoc analysis was planned for the printer, which was determined to determine the method statistically. To compare categorical protections is to use the Chi-square test. P < 0.05 will be considered future.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years or older
* Being diagnosed with lipedema according to Wold criteria
* Having type 1, 2 and 3 lipedema
* Having stage 1, 2 and 3 lipedema

Exclusion Criteria:

* Known rheumatic, endocrinological, neuromuscular, dermatological disease, kidney failure, liver failure and malignancy
* Having undergone surgery for lipedema
* Having poor circulation, open wound or infection in the lower extremities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Dual-energy X-ray absorptiometry (DXA) | measurements will be taken before treatment and at the 2nd week after treatment.
  DXA measurements were made with the patient in the supine position, with a radiation dose of 5.08 μSv, voltage 83.00 Kv, and current 0.2 mA from the head-to-heel distance by Osteosys Primus brand DXA device (Primus, X-ray densitometer, Osteosys Co. Ltd., Guro-gu, Seoul, Korea) will be made. With this measurement, the radiation dose received by the patient is very low and is below the daily natural radiation dose (7 μSv). With the obtained values, leg FM/total FM, android/gynoid fat ratios and fat mass (FM, fat mass) will be calculated using Osteosys Primus version 1.2.0 software. As a result of DXA measurements of the patients, Body Composition, Fat Mass, leg FM/total FM, Android/Gynoid FM values will be compared.
Volume measurement | measurements will be taken before treatment and at the 2nd week after treatment.
  For volume measurements in the lower extremities of the patients, circumference measurements will be taken from the ankle to the thigh at 4 cm intervals; then these values will be calculated automatically with the Pythagorean theorem in the Excel program.

SECONDARY OUTCOMES:
Quality of life - Nottingham Health Profile (NHP): | measurements will be taken before treatment and at the 2nd week after treatment.
  Nottingham Health Profile (NHP) is a general quality of life questionnaire that evaluates patients' perceptions of health problems and the effects of these problems on patients' activities of daily living. Pain, emotional reactions, sleep, social isolation, physical abilities and energy level subscales are evaluated. For each subscale, 0 points corresponds to the best health profile and 100 points corresponds to the worst health profile. The total NHP score is obtained by summing the subscale scores.
Algometric measurements | measurements will be taken before treatment and at the 2nd week after treatment.
  The pain threshold of the patients will be measured from the right and left extremities with a Wagner brand manual algometer. Before the evaluation is made, the patients will be informed about how the measurement will be made, and they will be asked to give information as soon as the feeling of pressure returns to the feeling of pain. For the measurement, the compression applied by keeping the probe of the algometer device perpendicular to the measuring surface will be gradually increased at the rate of approximately 0.5kg/cm²/s. The compression applied at the point where the patients feel pain will be terminated. The measurement will be made twice in the same area and 4 minutes will be waited before the second measurement is taken. The average of the two measurements will be recorded as the pressure pain threshold.
Visual Analogue Scale (VAS) | measurements will be taken before treatment and at the 2nd week after treatment.
  Pain intensity was measured with the Visual Analog Scale (0-10 mm; 0 means no pain, 10 means severe pain), which has a high reliability and validity in measuring musculoskeletal pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mihrinur Dilvin TÜRKÖZ, Study Director — Giresun University
Locations (1):
- Giresun University Training and Research Hospital, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aksoy H, Karadag AS, Wollina U. Cause and management of lipedema-associated pain. Dermatol Ther. 2021 Jan;34(1):e14364. doi: 10.1111/dth.14364. Epub 2020 Oct 12. PMID 33001552
- [Result] Fife CE, Maus EA, Carter MJ. Lipedema: a frequently misdiagnosed and misunderstood fatty deposition syndrome. Adv Skin Wound Care. 2010 Feb;23(2):81-92; quiz 93-4. doi: 10.1097/01.ASW.0000363503.92360.91. PMID 20087075
- [Result] Siems W, Grune T, Voss P, Brenke R. Anti-fibrosclerotic effects of shock wave therapy in lipedema and cellulite. Biofactors. 2005;24(1-4):275-82. doi: 10.1002/biof.5520240132. PMID 16403988
- [Result] Brandao ML, Soares HPDS, Andrade MDA, Faria ALSC, Pires RS. Efficacy of complex decongestive therapy for lymphedema of the lower limbs: a systematic review. J Vasc Bras. 2020 May 29;19:e20190074. doi: 10.1590/1677-5449.190074. PMID 34178058